CLINICAL TRIAL: NCT00988572
Title: Vestibular Rehabilitation for Patients With Fall-related Wrist Fractures - a Randomized Controlled Trial
Brief Title: Vestibular Rehabilitation for Patients With Fall-related Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Eva Ekvall Hansson, Associate professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Radius
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Wrist Fractures; Dizziness
Keywords: Wrist fractures; Vestibular asymmetry; Vestibular rehabilitation; Fall-related wrist fractures; Patients 50 years or older
MeSH Terms: conditions — Wrist Fractures; Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Vestibular rehabilitation, twice a week for 9 weeks
  Interventions: Other: Vestibular rehabilitation
- Control group (No Intervention): The patients in the control group does nothing, except for normal treatment for their wrist fracture.

INTERVENTIONS:
Other: Vestibular rehabilitation — The intervention program comprises of vestibular rehabilitation, at group sessions, twice a week for 9 weeks. The program is described in detail in table 1. Vestibular rehabilitation aims to facilitate rearrangement and recruitment of the control capacities of the vestibular system, by letting the patient be exposed to unstable body positions, such as standing on foam and performing head, trunk or eye-movements.
  Arms: Intervention group

SUMMARY:
Dizziness has been identified as a risk factor for fall and vestibular asymmetry has been found among patients with fall-related wrist fractures as well as among patients with hip-fracture. Since wrist fracture is a risk factor for hip-fracture, much effort is focused on preventing falls for risk-groups. Therefore, it would be interesting to find out if it is possible to influence vestibular asymmetry with vestibular rehabilitation.

The aim of this study is therefore to find out if vestibular rehabilitation can have any effect on vestibular function among patients with fall-related wrist fracture.

DETAILED DESCRIPTION:
Fall-related fractures are an increasing problem for the society. Almost 30% of persons over 65 years of age fall each year. In Sweden 627 persons out of 100 000 is treated in hospitals because of injury after a fall. In Malmö, the figure is 883 persons out of 100 000. However, not all falls lead to a fracture. Dizziness has been identified as a risk factor for fall and vestibular asymmetry has been found among patients with fall-related wrist fractures as well as among patients with hip-fracture.

Vestibular rehabilitation programs were first developed in the forties, originally used for peripheral vestibular disorder, in order to facilitate recovery. Modern research has widened the use of vestibular rehabilitation to patients with other causes of dizziness than peripheral vestibular disorders. Since wrist fracture is a risk factor for hip-fracture, much effort is focused on preventing falls for risk-groups. Therefore, it would be interesting to find out if it is possible to influence vestibular asymmetry with vestibular rehabilitation.

The aim of this study is therefore to find out if vestibular rehabilitation can have any effect on vestibular function among patients with fall-related wrist fracture.

ELIGIBILITY:
Inclusion Criteria:

* Fall-related wrist fracture
* 50 years or older

Exclusion Criteria:

* Younger than 50
* Wrist fracture not related to fall

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Vestibular function measured by head shake test | At baseline and at follow-up after 3 months

SECONDARY OUTCOMES:
Analyze of gait using electronic walkway | At baseline and at follow up after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Dep Clin Sci in Malmö/Family Practice, Malmo, Sweden

REFERENCES:
- [Background] Kristinsdottir EK, Jarnlo GB, Magnusson M. Asymmetric vestibular function in the elderly might be a significant contributor to hip fractures. Scand J Rehabil Med. 2000 Jun;32(2):56-60. doi: 10.1080/003655000750045550. PMID 10853718
- [Background] Kristinsdottir EK, Nordell E, Jarnlo GB, Tjader A, Thorngren KG, Magnusson M. Observation of vestibular asymmetry in a majority of patients over 50 years with fall-related wrist fractures. Acta Otolaryngol. 2001 Jun;121(4):481-5. PMID 11508508
- [Background] Hansson, EE. Vestibular Rehabilitation - for whom and how? Advances in Physiotherapy 9:106-116. 2007
- [Derived] Najafi DA, Dahlberg LE, Hansson EE. A combination of clinical balance measures and FRAX(R) to improve identification of high-risk fallers. BMC Geriatr. 2016 May 3;16:94. doi: 10.1186/s12877-016-0266-6. PMID 27142632